CLINICAL TRIAL: NCT01434524
Title: The Evaluation About the Prevention for the Development of Liver Tumorigenesis by the Oral Supplementation of Branched-chain Amino Acids
Brief Title: Prevention for the Development of Liver Tumorigenesis by the Oral Supplementation of Branched-chain Amino Acids
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kochi University (Other)
Responsible Party: Principal Investigator, Takehiro Okabayashi, Kochi Medical School, Kochi University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: LIVACT 0801; LIVACT 0801 (Other: Kochi Medical School)
Record Dates: First submitted 2011-09-13; First posted 2011-09-15 (Estimated); Last update posted 2011-09-15 (Estimated); Status verified 2011-09

CONDITIONS: Liver Cancer
MeSH Terms: conditions — Liver Neoplasms | interventions — Amino Acids, Branched-Chain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (No Intervention): normal dietary
- LIVACT (No Intervention): The present study used LIVACT for preoperative supplementation, commencing two weeks prior to surgery, and continuing for at least 6 months postoperatively with careful monitoring of compliance.
  Interventions: Drug: LIVACT

INTERVENTIONS:
Drug: LIVACT — LIVACT contains 13.0 g of free amino acids
  Other Names: branched-chain amino acid
  Arms: LIVACT

SUMMARY:
The long-term outcomes of branched-chain amino acid (BCAA) administration in patients undergoing hepatic resection remain unclear. The aim of this study is to assess the impact of oral supplementation with BCAA on the prevention for the development of liver tumorigenesis in patients undergoing liver resection.

DETAILED DESCRIPTION:
This study might demonstrate a tendency of the improvement in the cumulative tumor recurrence rate after hepatectomy for liver neoplasm in the Livact group compared to that in the Control Group. The investigators believe that BCAA seems to be a remarkable benefit for liver resection, especially on its reduction in the recurrence of liver cancer. This treatment regimen has potential to offer benefits for clinical use selectively, especially for patients with chronic liver diseases.

ELIGIBILITY:
Inclusion Criteria:

* These patients were scheduled for elective liver resection to treat hepatocellular carcinoma or adenocarcinoma of the liver.

Exclusion Criteria:

* a body-weight loss greater than 10% during the 6 months prior to surgery,
* the presence of distant metastases, or
* serious impairment of organ function due to respiratory, renal, or heart disease.

Ages: 16 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2007-04; Primary Completion 2008-10 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Postoperative tumor recurrence rate | 5 years follow up

SECONDARY OUTCOMES:
nutritional status | 5 years follow up
  The secondary endpoint was a comparison of measurements of body weight, arm muscle circumference (AMC) between patient groups.

CONTACTS AND LOCATIONS:
Overall Officials: Takehiro Okabayashi, MD, Principal Investigator — Kochi Medical School
Locations (1):
- Kochi Medical School, Nankoku, Kochi, Japan